CLINICAL TRIAL: NCT03909802
Title: Effect of Self- and Family Management of Diabetic Foot Ulcers Programs on Health Outcomes Among Individuals With Diabetic Foot Ulcers in Indonesia
Brief Title: Effect of Self- and Family Management of Diabetic Foot Ulcers Programs on Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Muhammadiyah Yogyakarta (Other)
Responsible Party: Principal Investigator, Sumarno Adi Subrata, PhD (Candidate), Principal investigator, Universitas Muhammadiyah Yogyakarta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRJ-2973 /LPDP.3/2016
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Diabete Mellitus; Diabetic Foot
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: The researcher will assess the obtained information relating to the patient having DFU and make a list of potentially eligible participants. Those who met the criteria will be random using research randomizer application. The participants will be provided an information sheet in the course of study objectives. Also, this objective will be informed to the owner of wound care clinics for improving the current treatment. Afterward, those who have a willingness to take part in this study will be interviewed to re-assess the eligible inclusion criteria. If they met with the criteria, they will be asked to sign informed consent, provide their home address and a convenient phone number as well. Prior to the study implementation, each eligible participant will be randomly assigned to determine whether he or she will be included either into an experimental or control group. This process will utilize a research randomizer application and the result will be protected by the researcher only.
Who Masked: Participant
Masking Description: The participants are masked from knowing the intervention given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): This arm will receive interventions consisting of self-management combined with family management programs.
  Interventions: Behavioral: Self-and family management of diabetic foot ulcers programs
- Control group (Placebo Comparator): Usual care refers to incorporating wound assessment, wound irrigation using NaCl, debridement, wound dressing, evaluation, and health education unmet with the self-and-family management of DFU program criteria in this study. All of the usual care will be performed and evaluated by the wound care nurses working at the selected clinics for this study.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Self-and family management of diabetic foot ulcers programs — The intervention combines self-management and family management focusing on behavioral changes in patients with diabetic foot ulcers. Self-management focuses on intensive health education of physical activities, diet, medication, foot care, and blood glucose control. Family management focuses on problem-solving, establishing roles, and effective involvement in providing care amid individuals suffering DFU.
  Arms: Experimental group
Other: Usual care — Usual care
  Arms: Control group

SUMMARY:
Brief description:

Diabetic foot ulcer (DFU) is described as a full-thickness lesion appearing at the skin of the foot along with infection, destruction of tissues due to neuropathy and/or peripheral artery disease (PAD) in people with diabetes (International Working Group on the Diabetic Foot, 2015). DFU commonly develops in middle-aged diabetic patients due to a long period of type 2 diabetes and poor adherence to control blood glucose level (Madanchi et al., 2013). Prevalence of DFU was four times higher than all combined cases of cancers in the world (Boulton, 2013; McInnes, 2012; Shaw, Sicree, & Zimmet, 2010). Numerous published studies have documented the rate of DFU at around 25% in Western Population (Boulton, 2013). Prevalence of DFU was stated between 7.3 % - 24 % at Indonesia hospitals (Soewondo, Ferrario, & Tahapary, 2013). An Indonesia nursing study recorded 12 % of diabetic foot ulcer cases from 249 individuals with type 2 diabetes in a regional hospital of Eastern Indonesia (Yusuf et al., 2015). Cases of infected DFU occurred in 98 patients in Sardjito Hospital Yogyakarta Indonesia in 2016 (Longdong, 2016).

In order to diminish the wide-reaching impact of DFU, a number of efforts have been performed in Indonesia. A study documented that sufficient diabetic patients' knowledge in performing foot care is able to decrease the incidence of DFU as well as LEA (Wulandini, Saputra, & Basri, 2013). Foot ulcers health education program was interrelated with patients' knowledge as well as attitudes concerning responsibility and involvement in DFU care (Arianti, Yetti, & Nasution, 2012; Mahfud, 2012; Sa'adah, Primanda, & Wardaningsih, 2016; Yoyoh, Mutaqqin, & Nurjanah, 2016). In line with their findings, another study confirmed that intensive health promotion increased patients' knowledge and practice in regard to perform routine foot care (Abbas, 2013). Also, health promotion intervention improves Hemoglobin A1c (HbA1c) in type 2 Diabetes (Brown, 1990; Norris, Lau, Smith, Schmid, & Engelgau, 2002; Florkowski, 2013). However, a number of these studies merely focused on the patient, not engaged family members as it may potentially reduce the effectiveness of therapy.

Accordingly, DFU is currently being a critical problems needs to be solved in Indonesia. Ensuring the engagement of both the patients and their families in treatment is an important strategy to deal with the chronic conditions (Baig, Benitez, Quinn, & Burnet, 2015; Miller & DiMatteo, 2013; Pamungkas, Chamroonsawasdi, & Vatanasomboon, 2017). Therefore, conducting a comprehensive intervention of DFU partnering individuals and their families in association with self-and family management is a groundbreaking and challenging strategy to overcome problems on DFU. We believe the findings of our study will render significant contributions to the national guideline of diabetes in Indonesia and prevention of LEA in nursing practice. Furthermore, it will be able to give promising results for accelerating DFU healing.

Purposes of the study:

The purpose of this study is to investigate the effect of a self- and family management of DFU programs on health outcomes as follows: behaviors (adherence to physical activities, medications, diet, foot care, and blood glucose control), family supports, biomarkers (HbA1c, wound size) in patients suffering DFU in Indonesia.

Hypothesis:

The study participants who joined completely the self- and family management of diabetic foot ulcer programs during three months would have a better behavior, biomarkers, and family supports than those who received the usual care.

DETAILED DESCRIPTION:
Study background:

Diabetic foot ulcer (DFU) is described as a full-thickness lesion appearing at the skin of the foot along with infection, destruction of tissues due to neuropathy and/or peripheral artery disease (PAD) in people with diabetes (International Working Group on the Diabetic Foot, 2015). DFU commonly develops in middle-aged diabetic patients due to a long period of type 2 diabetes and poor adherence to control blood glucose level (Madanchi et al., 2013). Prevalence of DFU was four times higher than all combined cases of cancers in the world (Boulton, 2013; McInnes, 2012; Shaw, Sicree, & Zimmet, 2010). Numerous published studies have documented the rate of DFU at around 25% in Western Population (Boulton, 2013). Prevalence of DFU was stated between 7.3 % - 24 % at Indonesia hospitals (Soewondo, Ferrario, & Tahapary, 2013). An Indonesia nursing study recorded 12 % of diabetic foot ulcer cases from 249 individuals with type 2 diabetes in a regional hospital of Eastern Indonesia (Yusuf et al., 2015). Cases of infected DFU occurred in 98 patients in Sardjito Hospital Yogyakarta Indonesia in 2016 (Longdong, 2016).

In long-term conditions, DFU leads to lower extremity amputation (LEA) (Pemayun, Naibaho, Novitasari, Amin, & Minuljo, 2016). Several factors relating to LEA were ischemia, neuropathy, end-stage renal disease, and depth of the wound along with infection (Widatalla, Mahadi, Shawer, Elsayem, & Ahmed, 2009). The incidence of LEA was forecasted to be more than a million per year (Peter-Riesch, 2016; Wu, Driver, Wrobel, & Armstrong, 2007). Two studies exposed that amputation procedures were performed every 20 seconds in the diabetic population in the world (Fejfarová et al., 2014). A recent study found the estimated range of amputations around 15 - 32 % in Indonesia (Soewondo et al., 2017). As a consequence, this condition will directly impact on the patient's health-related quality of life that encompasses physical, social, economic, and psychological aspects (Vileikyte, 2001).

In order to diminish the wide-reaching impact of DFU, a number of efforts have been performed in Indonesia. A study documented that sufficient diabetic patients' knowledge in performing foot care is able to decrease the incidence of DFU as well as LEA (Wulandini, Saputra, & Basri, 2013). Foot ulcers health education program was interrelated with patients' knowledge as well as attitudes concerning responsibility and involvement in DFU care (Arianti, Yetti, & Nasution, 2012; Mahfud, 2012; Sa'adah, Primanda, & Wardaningsih, 2016; Yoyoh, Mutaqqin, & Nurjanah, 2016). In line with their findings, another study confirmed that intensive health promotion increased patients' knowledge and practice in regard to perform routine foot care (Abbas, 2013). Also, health promotion intervention improves Hemoglobin A1c (HbA1c) in type 2 Diabetes (Brown, 1990; Norris, Lau, Smith, Schmid, & Engelgau, 2002; Florkowski, 2013). However, a number of these studies merely focused on the patient, not engaged family members as it may potentially reduce the effectiveness of therapy.

Currently, poor adherence to DFU treatment is taken into consideration on the diabetes population in Indonesia. Many diabetic patients had poor adherence in maintaining diabetes treatment which potentially leads to suboptimal diabetes outcomes involving increased blood glucose level, more hospital admissions, diabetes-related complications, and multiplied medical care costs (Putri, Yudianto, Kurniawan, & Titis, 2013; Waluya, 2008). To overcome this issue, intensive health promotion has been considered as the first-line approach in Indonesia (Windasari, 2014). In addition, strategies addressing poor adherence must be focused on reducing DFU complications in the future. This could be successfully achieved by incorporating family members in a particular intervention. A systematic review also pointed out that family support in a given treatment strengthens patient adherence to diabetes treatment (Rintala, Jaatinen, Paavilainen, & Astedt-Kurki, 2013). Efforts have been performed in Indonesia, even though it has some limitations. For instance, some studies merely addressed the age, gender, duration of diabetes and level of patient' education relating to the adherence, not focused on patients' motivation which is presently being the main problem in Indonesia (Ainni, 2017; Srikartika, Cahya, & Hardiati, 2016). Also, providing care to those suffering diabetes potentially becomes a burden on both physical and emotional aspects. Also, some individuals reported that they felt sadness when their family does not fully support their care. In line with these findings that, negative family support is the robust predictor for the patient's stress and decreased diabetes outcome (Pardamean & Dharmady, 2003; Isworo, Ekowati, Iskandar, & Latifah, 2018). The other study stated that patients receiving non-supportive care from a family member are more likely to have a poor blood glucose level (Isworo & Saryono, 2010). Moreover, the lack of family knowledge, low levels of self-efficacy, and insufficient social support from family members lead to poor diabetes self-management (Pamungkas, Chamroonsawasdi, & Vatanasomboon, 2017).

Due to the positive influence of family support on diabetes outcomes, the high-impact efforts to improve family support are considered to be necessary. Many studies described the family involvement in diabetes care consisting of providing emotional support, helping patients how to deal with diabetes problems, providing information and partnering in daily care. Nevertheless, they lacked information about how family members provide support in regard to self-management behaviors (Pamungkas, Chamroonsawasdi, & Vatanasomboon, 2017). As is well acknowledged, individuals' adherence along with family engagement to prescribed diabetes treatment is crucial to reach metabolic control lowering the complexities of diabetes, respectively. Family involvement in diabetes care may prevent patients from further complexities of diabetes (Isworo, Ekowati, Iskandar, & Latifah, 2018). Also, family members need to be informed in term of screening to prevent future complexities on individuals having diabetes, particular to those who have a sedentary lifestyle, a lack of physical activity, and an unhealthy diet (Soewondo, Ferrario, & Tahapary, 2013).

Managing individual with diabetes along with diabetic foot ulcers in the context of family management has been done by some researchers in Indonesia (Rahayu et al., 2014; Yusra, 2011; Prantika, Susilo, & Bagus, 2014; Putri et al., 2013; Sari, Susanti, & Sukmawati, 2014; Laily, 2016). As is culturally known in Indonesia, patients suffering diabetes live with their family which may either provide practical help in the management of diabetes or they were unsure to their abilities to help their family member particular in accidental situations. How family members respond will be different based upon their individual personalities, how committed they are to the individual with diabetes and their sense of responsibility (Budianto, 2015). Moreover, their reactions could indicate insufficient knowledge, fear, worried, or even a desire to support some help. For these reasons, addressing family engagement for those with diabetes is imperative since this is the context in which the majority of diabetes management happens. Family members play an essential role in a patient's disease management, incorporating them in self-care interventions may possibly render significant changes in patients' outcomes such as self-efficacy, perceived social support, diabetes knowledge, and diabetes self-care (Pamungkas, Chamroonsawasdi, & Vatanasomboon, 2017; Baig, Benitez, Quinn, & Burnet, 2015).

In Indonesia context, a study described that implementing a family management program (health education, motivational program, follow up care) during three months improved patients' quality of life and self-care (Rahayu et al., 2014; Yusra, 2011). The family management program is linked with the improvement of blood glucose control (Prantika, Susilo, & Bagus, 2014; Putri et al., 2013). Incorporating family members are helpful in diabetes therapy (Sari, Susanti, & Sukmawati, 2014). What's more, family dynamics have been indicated to have an impact on diabetes management in adults. Overall evidence above proofs a beneficial effect of a family role for people living with diabetes. However, partnership amid patients and their families in those study is lacking and the majority of individuals had insufficient knowledge in association with diabetic foot care which this condition may potentially increase the risk of LEA (Laily, 2016). Accordingly, family involvement in diabetes care is required to give the advantages to the individual outcomes such as patients' well-being, physical activities, medication adherence, routine blood glucose control, routine foot care and ability to maintain the changes to a healthier lifestyle. Also, intensive health education with respect to foot care strategies should be emphasized within the individuals and their families in Indonesia.

In 2015, PERKENI (Persatuan Endokrinologi Indonesia) or the Indonesian Society for Endocrinology, officially issued a national guideline of diabetes management entitled "konsensus pengelolaan dan pencegahan diabetes mellitus tipe 2 di Indonesia 2015" or consensus on management and prevention of type 2 diabetes in Indonesia 2015 (Persatuan Endokrinologi Indonesia, 2015). In this guideline, several approaches were recommended such as assessing illness trajectory, performing a physical examination, doing laboratory test (HbA1c only), implementing health education in lifestyle changing (diet and physical activities only), and using appropriate medication. Nevertheless, we have identified limitation to the guideline as follows: they have not specifically described the role of family involvement in the therapy. It stands to reason that family role is fundamental aspect due to their responsibility to address individuals' non-adherence to treatment at home. Also, several studies support that non-adherence to the diabetes treatment regimen is possibly the most common reason for poor health outcomes among individuals with diabetes in Indonesia (Putri, Yudianto, Kurniawan, & Titis, 2013; Waluya, 2008; Windasari, 2014). For that reason, the need to improve the guideline is essential as it would enhance the role of a family member in diabetes therapy along with preventing the further complications of DFU. Moreover, family-based interventions for individuals having diabetes have therefore proven to be an effective approach in improving treatment outcomes (Sanjari, Peyrovi, & Mehrdad, 2016). Another limitation discovered that guideline has not included wound size as a biomarker of evaluation in a given treatment. This marker is important to evaluate the progress of the DFU treatment (Roth-Albin et al., 2017; Alexiadou & Doupis, 2012).

Accordingly, DFU is currently being a critical problems needs to be solved in Indonesia. Ensuring the engagement of both the patients and their families in treatment is an important strategy to deal with the chronic conditions (Baig, Benitez, Quinn, & Burnet, 2015; Miller & DiMatteo, 2013; Pamungkas, Chamroonsawasdi, & Vatanasomboon, 2017). Therefore, conducting a comprehensive intervention of DFU partnering individuals and their families in association with self-and family management is a groundbreaking and challenging strategy to overcome problems on DFU. We believe the findings of our study will render significant contributions to the national guideline of diabetes in Indonesia and prevention of LEA in nursing practice. Furthermore, it will be able to give promising results for accelerating DFU healing.

Study objective:

The purpose of this study is to investigate the effect of a self- and family management of DFU programs on health outcomes as follows: behaviors (adherence to physical activities, medications, diet, foot care, and blood glucose control), family supports, biomarkers (HbA1c, wound size) in patients suffering DFU in Indonesia.

Study hypothesis:

The study participants who joined completely the self- and family management of diabetic foot ulcer programs during three months would have a better behavior, biomarkers, and family supports than those who received the usual care.

Study design:

A prospective, randomized controlled trial study proposes to investigate the effect of self- and family management of diabetic foot ulcers programs on health outcomes among individuals with diabetic foot ulcers in Indonesia. The self-and family management of DFU program was designed and adapted based upon a review of the literature along with Indonesia guideline of diabetes management developed by the Indonesian Society for Endocrinology (PERKENI). This study will be conducted during three months and data will be collected four times in the study implementation. HbA1c and wound size have been considered as the distal outcomes in this study. On the other hand, individual and family behavior known as the proximal outcomes will also be evaluated as the mediator of the distal outcomes.

The study will be put into operation in four phases, as follows: 1) pre-implementation program (O1, 05) consist of measuring several variables as baseline data: individual baseline data (behavior: adherence to physical activity, diet for diabetic patients, blood glucose control, and foot care; biomarkers: HbA1c and wound size); and family baseline data (family supports). 2) Implementing the program phase 1 and measuring individual and family behavior, wound size (X1). 3) Implementing the program phase 1 and measuring individual and family behavior, wound size (X2). 4) Implementing the program phase 1 and measuring individual and family behavior, and biomarkers (HbA1c and wound size) (X3). The study process was depicted in the chart below.

Program implementation:

Researcher preparation: prior to implementing the program, the researcher will prepare several elements such as participants characteristics obtained from selected wound care clinics. The procedure the usual care will also be assessed in this stage encompassing physical activity, medication, diet, foot care (i.e. wound care), and blood glucose control. Family management relating to DFU care will be collected from those clinics.

Program planning:

The self- and family management program of DFU was developed based upon the revised framework of self- and family management (Grey et al., 2015) and Konsensus Tatalaksana Diabetes Mellitus PERKENI Indonesia (2015). Additionally, the researcher added a literature review to improve the content of the guideline. In this study, the program will have two main outcomes consist of proximal outcome (family support and individual behavior) and distal outcomes (HbA1c and wound size). In this phase, the researcher will prepare the program-supported tools such as guideline from PERKENI and guideline developed by the researcher.

Self-management of DFU programs:

The self-management program will be implemented in one session within fifty minutes each session per week. However, it could be longer than as planned due to the atmosphere of discussion that possibly might change the duration. A total of 12 sessions was planned for program implementation. Teaching, group discussing, and counseling is the method that will be used during the study. On the following description, the contents of the self-management of DFU programs are presented.

Physical activities are critical for blood glucose management and overall health in individuals having diabetes. This includes all movement that increases energy use, whereas exercise is planned, structured physical activity. Regular physical activity may improve blood glucose control and reduces or prevent further complexities such as lower extremity amputations. In this session, participants will receive counseling, discussion, demonstration, and materials from the researcher. This material including the importance of performing physical activity according to the specific need of each individual with DFU. For instance, performing aerobic exercise (walking), weight training. Also, monitoring blood glucose before, during and many hours after activities to see how it effects on blood glucose levels.

Medication in diabetes refers to achieving optimal medication-taking behavior which is a collaborative process of communication and understanding between participants and the researcher. The objective of this phase is to improve medication-taking behavior in participants by modifying their approach on an individual such as discussion, assessment of the barrier to adhere to medications. Participants will be encouraged to taken multiple medications for hyperglycemia, diabetes-associated conditions, and other comorbidities. This approach associates with improved outcomes, including reduced complexities of DFU, re-admission to hospital, and fatality.

Diet goals for those suffering diabetes is to promote and support healthful eating patterns of diabetes, attain individualized glycemic, blood pressure, and lipid goals, achieve and maintain body weight goals, delay or prevent complications of diabetes, address individual nutrition needs based on personal and cultural preferences, maintain the pleasure of eating by providing positive messages about food choices, and provide the individual with diabetes with practical tools for day-to-day meal planning. In these sessions, the participant will be provided a discussion and counseling relating strategies to manage diet on diabetes and overcome the barrier that may interfere with the wound healing process.

Foot care (i.e. wound care) refers to regular to protect the foot from nerve damage, circulation problems, and infections that lead to serious diabetic foot problems. Preventing diabetes complications, possessing the risk factors, and having the ability to manage complications is part of a DFU self-management program. In this stage, the study participant will be encouraged to pay much attention to checking feet regularly, inspecting inside the shoes daily from foreign objects, keeping the feet clean and using moisturizer, cut nails regularly, and changing the wound dressing. Discussion and demonstration to perform wound care will also be conducted in this study.

Blood glucose control in this study refers to self-monitoring of blood glucose (SMBG) which is a crucial approach of diabetes therapy. SMBG has been recommended to attain a specific level of glycemic control and prevent acute hypoglycemia. The main goal of this phase is to collect detailed information about blood glucose levels at many time points to enable maintenance of a more constant glucose level by more precise regimens. Moreover, it can be used to aid in the adjustment of a therapeutic regimen in response to blood glucose values and to help individuals adjust their dietary intake, physical activity, and insulin doses to improve glycemic control on a day-to-day basis. Regular monitoring also enables tighter blood glucose control that diminish the long-term risks of diabetic complications. In Indonesia context, SMBG is the main concern of the individuals having diabetes that need to be improved by implementing this present study.

Family management of DFU programs:

Family management in this study focuses on three elements as follows the problem-solving discussion, establishing family roles in DFU care and effective involvement during DFU care. Family members come forward with understanding to deal with the condition alleviating the treatment burden as much as possible. For illustrative purposes, an individual having DFU always finds a family member for regular dressing and helping hand to handle daily activities. A family having patients with DFU should redistribute the roles of their members and show sensibility by managing inner conflicts, motivating the persons to adhere to treatment as per rule, and helping to nullify the worst impact of DFU. Motivational interviews, which can help to identify and reinforce the behavior change can be used to enhance the patient's motivation for diabetes self-care.

ELIGIBILITY:
Individual inclusion criteria:

1. Individual both men and women who were diagnosed stage 2 and more of DFU by certified wound care nurses.
2. Individual having DFU located on the one or two legs.
3. An individual who either regularly or not regularly visits the selected wound care clinics.
4. Individual not in the fasting period either in Ramadan or another occasion.
5. An individual who able to read and communicate in Indonesia language.

Individual exclusion criteria:

1. Individual who is hospitalized due to the complexities of diabetes.
2. Individual who at the end of life care.
3. Individual who is currently having any critical condition which potentially interferes data collection processes such as acute diabetic ketoacidosis and impaired consciousness.
4. An individual who has blindness due to diabetes or aging.

Family inclusion criteria:

1. The individual is the caregiver or family members of an individual having DFU.
2. An individual who able to read and communicate in Indonesia language.

Family exclusion criteria:

Individuals who attend the program less than 80 percent due to getting sick or other reasons.

Termination criteria:

This study will be suspended or terminated some or all research activities if events are identified representing serious or continuing noncompliance or unanticipated health issues involving risk to subjects or others related to DFU complications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-07-06 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-12-10 (Actual)

PRIMARY OUTCOMES:
HbA1c | up to 3 months
  Hemoglobin A1c (HbA1c) is defined as the glycated hemoglobin level that reflects the index of glycemia over 2-3 months. It is frequently used to examine glycemia in a patient with chronic diabetes. HbA1c will be measured by using a laboratory test examination certified by ISO 9001: 2015. After study accomplished, the expected goal of the HbA1c is less than 7 % as per recommendation by American Diabetes Association and Persatuan Endokrinologi Indonesia (American Diabetes Association, 2018; Persatuan Endokrinologi Indonesia, 2015). The measurement of this variable would be performed by a laboratory analyst.
Wound size | up to 3 months
  Wound size is defined as lesions of foot ulcers that can be quantitatively evaluated and categorized according to their length, width, and depth. In this study, wound size will be assessed throughout the study by implementing the photographic method as the gold standard measurement (Shetty et al., 2012). The PEDIS system will be used as a recommended classification (Game, 2016). This classification assesses perfusion (ischemia), extent (area), depth, infection, sensation (neuropathy). Individuals who have scored at < 7 is categorized at the low risk of the non-healing wound. Those who have > 7 are categorized at the high risk of a non-healing wound, amputation, and death (Chuan, Tang, Jiang, Zhou, & He, 2015). The stage of the wound would be assessed by a research assistant who is a certified wound care nurse.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Health Sciences, Universitas Muhammadiyah Magelang, Magelang, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No